CLINICAL TRIAL: NCT04044469
Title: Why Medical Reassurance Fails in Patients With Functional Somatic Symptoms - An Experimental Study on Cognitive Immunization
Brief Title: Reappraisal Of Medical Assurance (ROMA): An Experimental Study in Patients With Functional Somatic Symptoms
Acronym: ROMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Collaborators: University of Kaiserslautern-Landau (Other); Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: ROMA_199
Record Dates: First submitted 2019-07-16; First posted 2019-08-05 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2022-01

CONDITIONS: Somatic Symptom Disorder
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of three experimental groups in parallel for the duration of the study
Who Masked: Participant
Masking Description: The investigator randomly assigns participants to one of the experimental conditions. Participants are not aware which experimental condition they are allocated to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Immunization-enhancement (Experimental): This group receives an immunization-promoting manipulation aimed at triggering negative appraisals of the medical information received and questioning the validity of the medical reassurance. For this purpose, a standardized information text is presented to the participants after receipt of the doctor's report, in which it is stated that the standard medical diagnosis in gastroenterology is often not particularly accurate and that serious diseases are from times to times overlooked. As a further factor contributing to the non-detection of diseases, it is mentioned that doctors are often under time pressure and thus do not have sufficient time to ask patients for all important information. It is believed that communicating this information will result in participants continuing to report high probabilities of serious illness despite the previously received findings report.
  Interventions: Behavioral: Immunization-enhancement
- Immunization-inhibition (Experimental): The aim of the immunization-inhibiting manipulation is to increase the probability that the normal test results obtained will be used to reduce worries about a serious illness. The participants of this group receive - analogous to the immunization-promoting group - a standardized information text which states that the standard medical diagnosis in gastroenterology is very accurate and that the physicians are very often correct in their initial diagnostic assessment, especially with regard to the assessment of a serious organic disease. This is supported by two scientific publications. The aim of this information is to increase the value of the results obtained, so that the participants are more reassured as a result of the inconspicuous test results and use them to correct their health-related concerns.
  Interventions: Behavioral: Immunization-inhibition
- Control group (Experimental): This group does not receive additional information after the doctor's report.
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: Immunization-enhancement — This group receives a standardized information text, suggesting that medical diagnostics is not very accurate. Reasons for why a serious disease is overlooked are mentioned and discussed.
  Arms: Immunization-enhancement
Behavioral: Immunization-inhibition — This group receives a standardized information text, suggesting that medical diagnostics is very accurate and that doctors are very often right in their first initial diagnostic assessments.
  Arms: Immunization-inhibition
Behavioral: Control group — This group receives no further information after watching the videotaped doctor's report.
  Arms: Control group

SUMMARY:
Research has shown that patients with functional somatic symptoms continue to worry about having a serious disease despite medical reassurance from their doctors. This study aims to investigate whether cognitive immunization is a mechanism that underlies the sustained concern about having serious disease. To this end, the use of cognitive immunization strategies will be experimentally modulated after receipt of medical test results.

DETAILED DESCRIPTION:
It is known from research on functional somatic symptoms that patients continue to worry about having a serious illness despite receiving medical reassurance and normal medical test results. However, the psychological mechanisms underlying this maintenance of concern are largely unknown. The planned study will therefore apply knowledge from depression research to this question: In the field of depression there is sound evidence that people with depressive symptoms maintain negative expectations despite positive experiences to the contrary, and in previous work it was shown that this is due to a cognitive re-appraisal of expectation-disconfirming experiences, referred to as cognitive immunization. The planned study seeks to investigate whether cognitive immunization is also a mechanism underlying sustained concerns about having a serious disease despite medical reassurance in patients with functional somatic symptoms. For this purpose, participants are presented with a vignette in which gastrointestinal complaints are reported; participants are instructed to imagine to suffer from these symptoms and to go a doctor to have their symptoms examined. Subsequently, participants watch a videotaped doctor's report in which a family doctor discusses the results of several medical tests that have been carried out to exclude the possibility of some serious diseases, such as colon cancer. In this report, the doctor states clearly that, based on the test results, a serious disease is very unlikely. Afterwards, participants of some experimental groups receive additional information on the accuracy of medical diagnostics, aimed at differentially varying the appraisal of the medical reassurance received.

The experimental conditions described above apply only to the sample of patients with functional somatic symptoms (inclusion and exclusion criteria see below). In addition, we will also recruit a clinical (patients with depression, n=30) and healthy control group (n=30). These control groups will not undergo the cognitive immunization manipulation, but will only pass through the basic procedure of the experimental paradigm, that is, the same procedure as the control group from the sample of patients with functional somatic symptoms. These two control groups (healthy and clinical) are recruited to replicate previous findings showing that patients with somatic symptoms report increased probabilities of suffering from a serious disease compared to patients with depression and healthy control participants. Below, we will only present the inclusion and exclusion criteria of the sample with functional somatic symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of a somatoform disorder (F45.x) (as assessed with the SKID interview)
* Age between 18 and 69
* Sufficient German language skills

Exclusion Criteria:

* acute life-threatening disease
* diagnosed mental disorder other than the somatoform disorder that is considered the primary diagnosis (people with other comorbid mental disorders are not excluded if the somatoform disorder is the primary diagnosis)

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-10-23 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2021-12-23 (Actual)

PRIMARY OUTCOMES:
Likelihood of a serious disease scale | 2 minutes after the doctor's report
  Numerical analogue scale to assess the likelihood of having a serious disease (0 = serious disease excluded; 100 = serious disease for sure)

SECONDARY OUTCOMES:
Cognitive immunization against medical reassurance scale | 5 minutes after the doctor's report
  Assessment of cognitive reappraisal of medical reassurance; each item is scored 1-7 (1 = totally disagree; 7 = totally agree)

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Kube, PhD, Principal Investigator — University of Kaiserslautern-Landau
Locations (1):
- University of Koblenz-Landau, Landau, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kube T, Riecke J, Heider J, Ballou SK, Glombiewski JA, Rief W, Barsky AJ. How the integration of normal medical test results can be improved in patients with somatoform disorders-An experimental study. Health Psychol. 2023 Feb;42(2):103-112. doi: 10.1037/hea0001243. Epub 2022 Dec 22. PMID 36548078